

### ClinicalTrials.gov Protocol Registration and Results System (PRS) Receipt

Release Date: October 19, 2020

### ClinicalTrials.gov ID: [Not yet assigned]

# **Study Identification**

Unique Protocol ID: CMUH109-REC2-131

Brief Title: The Effectiveness of Acupressure for Managing Postoperative Pain and Anxiety

in Patients With Thoracoscopic Surgery.

Official Title: Professor, School of Nursing, China Medical University Hospital, Principal

Investigator.

Secondary IDs:

# **Study Status**

Record Verification: October 2020

Overall Status: Recruiting

Study Start: September 20, 2020 [Actual]

Primary Completion: August 2021 [Anticipated]

Study Completion: September 2021 [Anticipated]

# Sponsor/Collaborators

Sponsor: Wei-Fen Ma

Responsible Party: Sponsor-Investigator

Investigator: Wei-Fen Ma [Ihdaisy]

Official Title: Professor, School of Nursing Affiliation: China Medical University Hospital

Collaborators: China Medical University Hospital

# **Oversight**

U.S. FDA-regulated Drug: No

U.S. FDA-regulated Device: No

U.S. FDA IND/IDE: No

Human Subjects Review: Board Status: Approved

Approval Number: CMUH109-REC2-131

Board Name: Research Ethics Committee China Medical University and

Hospital, Taichung, Taiwan

Board Affiliation: China Medical University and Hospital

Phone: 886-4-22052121

Email: Address: 2 Yude Road, Taichung, 40447, Taiwan

Data Monitoring: No FDA Regulated Intervention: No

# **Study Description**

Brief Summary: The purpose of this study is to explore the effectiveness of acupressure

for managing postoperative pain, anxiety, analgesia consumption, early

ambulation, and comfort in patients with thoracoscopic surgery.

Detailed Description: Thoracoscopic surgery is the surgical used to removal of a section or a

segment of a lung lobe. One US national survey reported that 80% of patients undergoing pulmonary surgery experienced acute pain. 75-86% of these patients pointed out that experienced moderate, severe, or extreme pain, especially, on the 1st day after thoracoscopic surgery. However, inappropriate pain management after surgery is associated with limited the healing process, increased workload of heart, prolonged pulmonary rehabilitation, and increased medical costs, and can be a prediction of developing chronic pain. Acupressure is a nonpharmacological treatment for the management of postoperative pain. Recent studies have found that the application of acupressure is effective in decreasing operative pain intensity, morphine related side effects, and opioid consumptions after surgery. However, there was no further research about the

role of acupressure applied to thoracoscopic surgery.

## **Conditions**

Conditions: Lung Diseases

Keywords: acupressure

thoracoscopic surgery

acute pain anxiety comfort

# **Study Design**

Study Type: Interventional

Primary Purpose: Supportive Care

Study Phase: N/A

Interventional Study Model: Parallel Assignment

Number of Arms: 2

Masking: Single (Participant)

Allocation: Randomized

Enrollment: 200 [Anticipated]

### Arms and Interventions

| Arms | Assigned Interventions |
|---|---|
| Experimental: acupressure | acupressure |
| After recruitment, participants will be randomized | The acupressure involves the "Vaccaria Semen" |
| to receive acupressure or control group. In the | within skin-colored adhesive tape that placed on |

| Arms | Assigned Interventions |
|---|---|
| acupressure group, participants will receive acupressure treatment. | the "Neiguan" and "Shenmen" acupoints as an intervention measure. Continue to massage the acupoints with fingertips for 10 minutes, 3 times per day (8 and 12 in the morning, and 4 in the afternoon). The adhesive tape will be retained in situ for 2 days. |
| No Intervention: routine care After recruitment, participants will be randomized to receive acupressure or control group. In the control group, participants will receive routine care, including routine pain control. | |

### **Outcome Measures**

## Primary Outcome Measure:

1. Pain:Changes from baseline pain scale at post-operative day 2, after intervention. as assessed by Visual Analogue Scale-Pain (VAS-P). The VAS#P scale is comprised of a horizontal line 100mm long with the indication "no pain" to the left and "worst possible pain" to the right. possible scores varied between 0–100. A higher scores mean a worse outcome.

[Time Frame: Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 8 ante meridiem (AM), before intervention; post-operative day 1, 5 PM, after intervention; and post-operative day 2, 5 PM, after intervention]

### Secondary Outcome Measure:

#### 2. Anxiety

as assessed by Visual Analogue Scale-Anxiety(VAS-A). The VAS#A scale is comprised of a horizontal line 100mm long with the indication "no anxiety" to the left and "worst possible anxiety" to the right. possible scores varied between 0–100. A higher scores mean a worse outcome.

[Time Frame: Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 9 ante meridiem (AM), before intervention; post-operative day 1, 5 PM, after intervention; and post-operative day 2, 5 PM, after intervention.]

#### 3. Anxiety

as assessed by State-Trait Anxiety Inventory (STAI) Y form (STAI-Y1). It is 20 questions, which were rated from 1–4. Possible scores varied between 20–80. A STAI-Y1 score>40 as evidence of a state of anxiety.

[Time Frame: Time Frame: Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 8 ante meridiem (AM), before intervention; and post-operative day 2, post meridiem (PM), after intervention.]

### Other Pre-specified Outcome Measures:

## 4. Analgesia Consumption

Injection time of morphine and ketorolac would be recorded.

[Time Frame: during the whole admission, an average of 4 day.]

#### 5. Comfort

as assessed by Shortened General Comfort Questionnaire

[Time Frame: Measure at before operation day,7 post meridiem (PM), before operation; post-operative day 1, 8 ante meridiem (AM), before intervention; and post-operative day 2, 5pm, after intervention]

#### 6. Heart rate variability

as assessed by Nexus-10, wireless Biofeedback/Neurofeedback system

[Time Frame: Measure at before operation day, 7 post meridiem (PM), before operation; post-operative day1, 8 ante meridiem (PM), before intervention; post-operative day 1, 5 post meridiem (PM), after intervention; and post-operative day 2, 5 PM, after intervention.]

### 7. Early ambulation

The first ambulation time: act to walk with or without any kind of assistant after operation.

# **Eligibility**

Minimum Age: 20 Years

Maximum Age:

Sex: All

Gender Based:

Accepts Healthy Volunteers: Yes

Criteria: Inclusion Criteria:

- pulmonary lung disease and will be scheduled to undergo a thoracoscopic wedge resection, segmentectomy, or lobectomy.
- American Society of Anesthesiologist physical status of Classes I-II,
- · both forearms without missing limbs or arteriovenous fistula
- · ability to communicate in Taiwanese or Chinese, and
- · agreement to participate in this study.

#### **Exclusion Criteria:**

- diagnosed as malignant neoplasm with lung meta,
- · Had a stroke or peripheral vascular disease
- Platelet count less than 20 x 10^3/mm^3
- · Using the patient controlled analgesia, and
- any known mental illness or memory dysfunction.

#### Contacts/Locations

Central Contact Person: Wei-Fen Ma, Ph.D

Telephone: 04-22053366 Ext. 7107 Email: Ihdaisy@mail.cmu.edu.tw

Central Contact Backup: Wei-Fen Ma, Ph.D

Study Officials: Wei-Fen Ma, Ph.D

Study Principal Investigator China Medical University, China

Locations: Taiwan

China Medical University

[Recruiting]

Taichung, Taiwan, 40447

Contact: Wei-Fen Ma, PHD 04-22053366 Ext. 7107

Ihdaisy@mail.cmu.edu.tw

Contact: Wei-Fen Ma, PHD 04-22053366 Ext. 7107 Ihdaisy@gmail.com

Principal Investigator: Wei-Fen Ma, Ph.D Sub-Investigator: Hsing-Chi Hsu, MSc

# **IPDSharing**

Plan to Share IPD: No

#### References

Citations: **[Study Results]** Abouarab AA, Rahouma M, Kamel M, Ghaly G, Mohamed A. Single Versus Multi-Incisional Video-Assisted Thoracic Surgery: A Systematic Review and Meta-analysis. J Laparoendosc Adv Surg Tech A. 2018 Feb;28(2):174-185. doi: 10.1089/lap.2017.0446. Epub 2017 Nov 6. Review. PubMed 29106318

Amico, T. A. D. (2007). Thoracoscopic Lobectomy. Journal of Medical Sciences, 27(3), 95-100. https://doi.org/10.6136/JMS.2007.27(3).095

Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-40, table of contents. PubMed 12873949

Au DW, Tsang HW, Ling PP, Leung CH, Ip PK, Cheung WM. Effects of acupressure on anxiety: a systematic review and meta-analysis. Acupunct Med. 2015 Oct;33(5):353-9. doi: 10.1136/acupmed-2014-010720. Epub 2015 May 22. PubMed 26002571

Batvani M, Yousefi H, Valiani M, Shahabi J, Mardanparvar H. The Effect of Acupressure on Physiological Parameters of Myocardial Infarction Patients: A Randomized Clinical Trial. Iran J Nurs Midwifery Res. 2018 MarApr;23(2):143-148. doi: 10.4103/ijnmr.IJNMR 83 16. PubMed 29628963

Boker A, Brownell L, Donen N. The Amsterdam preoperative anxiety and information scale provides a simple and reliable measure of preoperative anxiety. Can J Anaesth. 2002 Oct;49(8):792-8. PubMed 12374706

Chang LH, Hsu CH, Jong GP, Ho S, Tsay SL, Lin KC. Auricular acupressure for managing postoperative pain and knee motion in patients with total knee replacement: a randomized sham control study. Evid Based Complement Alternat Med. 2012;2012:528452. doi: 10.1155/2012/528452. Epub 2012 Jul 10. PubMed 22844334

Chang S. The meridian system and mechanism of acupuncture: a comparative review. Part 3: Mechanisms of acupuncture therapies. Taiwan J Obstet Gynecol. 2013 Jun;52(2):171-84. doi: 10.1016/j.tjog.2013.04.005. Review. PubMed 23915848

Chang S. The meridian system and mechanism of acupuncture-a comparative review. Part 1: the meridian system. Taiwan J Obstet Gynecol. 2012 Dec;51(4):506-14. doi: 10.1016/j.tjog.2012.09.004. Review. PubMed 23276552

Chen JS, Cheng YJ, Hung MH, Tseng YD, Chen KC, Lee YC. Nonintubated thoracoscopic lobectomy for lung cancer. Ann Surg. 2011 Dec;254(6):1038-43. doi: 10.1097/SLA.0b013e31822ed19b. PubMed 21869676

Chen T, Wang K, Xu J, Ma W, Zhou J. Electroacupuncture Reduces Postoperative Pain and Analgesic Consumption in Patients Undergoing Thoracic Surgery: A Randomized Study. Evid Based Complement Alternat Med. 2016;2016:2126416. doi: 10.1155/2016/2126416. Epub 2016 Mar 17. PubMed 27073400

Coutaux A. Non-pharmacological treatments for pain relief: TENS and acupuncture. Joint Bone Spine. 2017 Dec;84(6):657-661. doi: 10.1016/j.jbspin.2017.02.005. Epub 2017 Feb 20. Review. PubMed 28219657

Danoff JR, Goel R, Sutton R, Maltenfort MG, Austin MS. How Much Pain Is Significant? Defining the Minimal Clinically Important Difference for the Visual Analog Scale for Pain After Total Joint Arthroplasty. J Arthroplasty. 2018 Jul;33(7S):S71-S75.e2. doi: 10.1016/j.arth.2018.02.029. Epub 2018 Feb 22. PubMed 29567002

Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. PubMed 8598068

Endler NS, Kocovski NL. State and trait anxiety revisited. J Anxiety Disord. 2001 May-Jun;15(3):231-45. Review. PubMed 11442141

Engen DJ, Carns PE, Allen MS, Bauer BA, Loehrer LL, Cha SS, Chartrand CM, Eggler EJ, Cutshall SM, Wahner-Roedler DL. Evaluating efficacy and feasibility of transcutaneous electrical nerve stimulation for postoperative pain after video-assisted thoracoscopic surgery: A randomized pilot trial. Complement Ther Clin Pract. 2016 May;23:141-8. doi: 10.1016/j.ctcp.2015.04.002. Epub 2015 Apr 20. PubMed 25935320

Erdogan M, Erdogan A, Erbil N, Karakaya HK, Demircan A. Prospective, Randomized, Placebo-controlled Study of the Effect of TENS on postthoracotomy pain and pulmonary function. World J Surg. 2005 Dec;29(12):1563-70. PubMed 16331341

Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. Review. PubMed 24829420

Frödin, M., & Warrén Stomberg, M. (2014). Pain management after lung surgery. Nursing Reports, 4(1). https://doi.org/10.4081/nursrep.2014.3225

Fu, J., & Yang, M. (2019). The Yellow Emperor's Classic of Medicine — Essential Questions: Translation of Huangdi Neijing Suwen. WORLD SCIENTIFIC. https://doi.org/10.1142/11080

Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/ JPR.S144066. eCollection 2017. Review. PubMed 29026331

Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. Review. PubMed 24237004

Gupta A, Kaur K, Sharma S, Goyal S, Arora S, Murthy RS. Clinical aspects of acute post-operative pain management & its assessment. J Adv Pharm Technol Res. 2010 Apr;1(2):97-108. PubMed 22247838

Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. Review. PubMed 22588748

Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. PubMed 1071419

Hsiung DY, Liu CW, Cheng PC, Ma WF. Using non-invasive assessment methods to predict the risk of metabolic syndrome. Appl Nurs Res. 2015 May;28(2):72-7. doi: 10.1016/j.apnr.2014.12.001. Epub 2014 Dec 17. PubMed 25908541

Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. PubMed 4139420

Kaplowitz J, Papadakos PJ. Acute pain management for video-assisted thoracoscopic surgery: an update. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):312-21. doi: 10.1053/j.jvca.2011.04.010. Epub 2011 Jun 25. Review. PubMed 21705236

Kibler VA, Hayes RM, Johnson DE, Anderson LW, Just SL, Wells NL. Cultivating quality: early postoperative ambulation: back to basics. Am J Nurs. 2012 Apr;112(4):63-9. doi: 10.1097/01.NAJ.0000413460.45487.ea. PubMed 22456575

Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. PubMed 10702461

Kolcaba K, Schirm V, Steiner R. Effects of hand massage on comfort of nursing home residents. Geriatr Nurs. 2006 Mar-Apr;27(2):85-91. PubMed 16638478

Kuroda H, Mizuno H, Dejima H, Watanabe K, Yoshida T, Naito Y, Sakao Y. A retrospective study on analgesic requirements for thoracoscopic surgery postoperative pain. J Pain Res. 2017 Nov 15;10:2643-2648. doi: 10.2147/JPR.S147691. eCollection 2017. PubMed 29180890

Ma WF, Liu YC, Chen YF, Lane HY, Lai TJ, Huang LC. Evaluation of psychometric properties of the Chinese Mandarin version State-Trait Anxiety Inventory Y form in Taiwanese outpatients with anxiety disorders. J Psychiatr Ment Health Nurs. 2013 Aug;20(6):499-507. doi: 10.1111/j.1365-2850.2012.01945.x. Epub 2012 Jul 5. PubMed 22762356

Mehta P, Dhapte V, Kadam S, Dhapte V. Contemporary acupressure therapy: Adroit cure for painless recovery of therapeutic ailments. J Tradit Complement Med. 2016 Jul 22;7(2):251-263. doi: 10.1016/j.jtcme.2016.06.004. eCollection 2017 Apr. Review. PubMed 28417094

Nomori H, Horio H, Naruke T, Suemasu K. What is the advantage of a thoracoscopic lobectomy over a limited thoracotomy procedure for lung cancer surgery? Ann Thorac Surg. 2001 Sep;72(3):879-84. PubMed 11565674

Pogatzki-Zahn EM, Segelcke D, Schug SA. Postoperative pain-from mechanisms to treatment. Pain Rep. 2017 Mar 15;2(2):e588. doi: 10.1097/PR9.000000000000588. eCollection 2017 Mar. PubMed 29392204

Sharifi Rizi M, Shamsalinia A, Ghaffari F, Keyhanian S, Naderi Nabi B. The effect of acupressure on pain, anxiety, and the physiological indexes of patients with cancer undergoing bone marrow biopsy. Complement Ther Clin Pract. 2017 Nov;29:136-141. doi: 10.1016/j.ctcp.2017.09.002. Epub 2017 Sep 5. PubMed 29122251

Tamura M, Shimizu Y, Hashizume Y. Pain following thoracoscopic surgery: retrospective analysis between single-incision and three-port video-assisted thoracoscopic surgery. J Cardiothorac Surg. 2013 Jun 12;8:153. doi: 10.1186/1749-8090-8-153. PubMed 23759173

Wang Y, Tang H, Guo Q, Liu J, Liu X, Luo J, Yang W. Effects of Intravenous Patient-Controlled Sufentanil Analgesia and Music Therapy on Pain and Hemodynamics After Surgery for Lung Cancer: A Randomized Parallel Study. J Altern Complement Med. 2015 Nov;21(11):667-72. doi: 10.1089/acm.2014.0310. Epub 2015 Sep 2. PubMed 26331434

You WY, Yeh TP, Lee KC, Ma WF. A Preliminary Study of the Comfort in Patients with Leukemia Staying in a Positive Pressure Isolation Room. Int J Environ Res Public Health. 2020 May 22;17(10). pii: E3655. doi: 10.3390/ijerph17103655. PubMed 32456113

Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. Review. PubMed 21704871

Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. Review. PubMed 21704871

World Health Organization. (1991). A Proposed Standard International Acupuncture Nomenclature: Report of a WHO Scientific Group. Annals of Internal Medicine, 115(4), 335. https://doi.org/10.7326/0003-4819-115-4-335\_2

Links: URL: https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system

Description American Society of Anesthesiologists Physical Status

Classification System.

### Available IPD/Information:

U.S. National Library of Medicine | U.S. National Institutes of Health | U.S. Department of Health & Human Services

Cover page

Official title: China Medical University Hospital

NCT number: NCT04595253

Title: The Effectiveness of Acupressure for Managing Postoperative Pain and

Anxiety in Patients With Thoracoscopic Surgery

**Statistical Analysis Plan** 

SPSS statistical software was used for data analysis, independent t test

and chi-square test were used for descriptive analysis. A mixed model

with repeated analysis was used to examine the effect of acupressure on

pain, anxiety, and comfort. Regression analysis was to explore the

influences of pain, anxiety, and comfort for study patients with

thoracoscopic Surgery.

**Primary Completion Date** 

The patient experienced moderate pain and anxiety after thoracoscopic

significant difference in demographic surgery. There was no

characteristics between the two groups before they received surgery.

The experimental group, compared with the control group, pain intensity

(p<0.01) and anxiety score (p<0.05) were statistically significant lower on

day 1 and day 2 after intervention. The STAI-Y1 score (F=2.514, p=.086)

and comfort level (F=2.953, p=.057) were no significant differences after

intervention between two groups. The longer intervention, the

significantly decreased pain intensity (p<0.05) for surgical procedures

with lighter pain perception.